CLINICAL TRIAL: NCT02009085
Title: Pilot Study to Asses the Identification of Melanoma in Skin Lesions.
Brief Title: Pilot Study to Determine Feasibility of Benign and Malignant Skin Lesion Detection.
Status: Completed | Type: Observational
Sponsor: Orlucent, Inc (Industry)
Collaborators: Clalit Health Services (Other)
Responsible Party: Sponsor
Other Study IDs: KH 2012
Record Dates: First submitted 2013-11-25; First posted 2013-12-11 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Skin Lesions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Individuals undergoing skin excision.: Skin lesions are under suspicion for skin cancer.

SUMMARY:
In this study a fluorescent contrast dye is applied to a suspicious skin lesion.

Images are acquired and processed. The information is used to develop a prediction model for the presence of malignant transformation in the skin.

DETAILED DESCRIPTION:
Images acquired in the study are used for the development of a software analysis program.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Individual is scheduled for a skin biopsy in toto
* The lesion is pigmented or non pigmented
* Lesions may be under suspicion for basal cell carcinoma, squamous cell carcinoma, actinic keratosis, nevi, melanoma, seborrheic keratosis.
* The lesion is accessible to the imaging device

Exclusion Criteria:

* The patient has sensitive skin and easily breaks out in rash
* The lesion is within 1 cm of the eye
* The lesion is on mucosal surfaces (e.g., lips, genitals)
* Pregnant females
* Taking medications that pigments the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients above 18 years scheduled for a skin biopsy.
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2013-06; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Correlation between imaging and pathology. | No long term follow up is necessary.
  Patients are imaged and then undergo a biopsy. Images are used to develop a software predicting model based on pathology. Sensitivity and specificity parameters are calculated.
  No long term follow up is required since the biopsy is performed on the skin imaged. The follow up required is for the pathology for the skin excised.

SECONDARY OUTCOMES:
Acute response | up to 1 day
  The acute dermal response to the imaging procedure is evaluated.

OTHER OUTCOMES:
None specified. | 0
  no other outcome is specified in the .

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Ullmann, MD, Principal Investigator — Rambam Health Care Campus